CLINICAL TRIAL: NCT00400062
Title: MIND-ICU Study: Delirium and Dementia in Veterans Surviving ICU Care
Status: Completed | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Vanderbilt University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: MHBB-022-06S
Record Dates: First submitted 2006-11-15; First posted 2006-11-16 (Estimated); Last update posted 2019-04-19 (Actual); Status verified 2019-04

CONDITIONS: Delirium; Aging; Dementia
Keywords: Critical care; delirium; long-term cognitive impairment; mechanical ventilation; critical illness; dementia; aging; sedatives and analgesics
MeSH Terms: conditions — Delirium; Dementia; Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ICU survivors: The investigators will measure the independent contribution of risk factors such as delirium and exposure to sedative and analgesic medications to the incidence of long-term CI.

SUMMARY:
This will be the first large cohort study to define the epidemiology of and identify modifiable risk factors for long-term CI and functional deficits of ICU survivors. The investigators will measure the independent contribution of risk factors such as delirium and exposure to sedative and analgesic medications to the incidence of long-term CI, controlling for established risk factors (e.g., age, pre-existing CI, and apoE genotype). Defining the contributions of these risk factors will make it possible to develop preventive and/or treatment strategies to reduce the incidence, severity and/or duration of long-term CI and improve functional recovery of patients with acute critical illness.

DETAILED DESCRIPTION:
Advances in critical care have led to improved survival among those admitted to intensive care units (ICUs). However, survival is lower among those who develop ICU delirium, and the quality of life among survivors may be affected by post-ICU long-term cognitive impairment (CI) that lasts months to years. Long-term CI has been studied predominantly following cardiopulmonary bypass. In the much larger group of medical and general surgical ICU patients, the extent of this problem and its relationship to health-related quality of life is poorly characterized. Evidence from 6 pilot cohorts (including the investigators') totaling ~300 patients suggests that an astonishing 30% to 80% of ICU survivors experience long-term CI functionally equivalent to mild/moderate dementia although it may not be progressive (and thus will be referred to as long-term CI). Interestingly, this cognitive impairment arises independent of severity of illness, and older patients appear particularly prone. The investigators' work and the work of others have shown that delirium is a major independent risk factor for impaired cognitive function at hospital discharge and increased mortality at 6 months. While it is not clear whether delirium itself is injurious to the brain or is simply a marker of brain injury, it is clear that the onset of delirium in the ICU should not be considered innocuous; rather, it may be a determinant of long-term CI and health-related quality of life. Having spent the last 8 years studying delirium and drug exposure during acute phases of critical illness and long-term CI after hospitalization, the investigators are thoroughly prepared to continue the next phases of investigation in VA (Department of Veterans Affairs) patients, many of whom are older and disproportionately at risk for adverse outcomes following ICU care.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be included if they are adult patients in a medical and/or surgical ICU receiving treatment for any of the following: respiratory failure or cardiogenic or septic shock.

Exclusion Criteria:

Patients who meet the inclusion criteria will be excluded if they meet any of the following criteria:

* Cumulative ICU time > 5 days in the past 30 days, not including the current ICU stay, as this might create a state of flux regarding patients' cognitive baseline.
* Severe cognitive or neurodegenerative diseases that prevent a patient from living independently at baseline, including mental illness requiring institutionalization, acquired or congenital mental retardation, known brain lesions, traumatic brain injury, cerebrovascular accidents with resultant moderate to severe cognitive deficits or ADL dependency, Parkinson's disease, Huntington's disease, severe Alzheimer's disease or dementia of any etiology.
* ICU admission post cardiopulmonary resuscitation with suspected anoxic injury
* An active substance abuse or psychotic disorder, or a recent (within the past 6 months) serious suicidal gesture necessitating hospitalization. This exclusion that will enrich follow-up rates by avoiding patients with whom it is particularly challenging to maintain long-term contact.
* Blind, deaf, or unable to speak English, as these conditions would preclude our ability to perform the follow-up evaluation interviews.
* Overly moribund and not expected to survive for an additional 24 hours and/or withdrawing life support to focus on comfort measures only.
* Prisoners.
* Patients who live further than 200 miles from the study site and who do not regularly visit the study site area.
* The onset of the current episode of respiratory failure, cardiogenic shock, or septic shock was >72 hours ago.
* Patients who have had cardiac bypass surgery within the past 3 months (including the current hospitalization).
* Patients who are homeless and have no secondary contact person available. This exclusion will enrich follow-up rates by avoiding patients with whom it is particularly challenging to maintain long-term contact.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Medical and Surgical ICUs
Sampling Method: Probability Sample
Enrollment: 800 (Actual)
Dates: Start 2007-07-01 (Actual); Primary Completion 2010-12-01 (Actual); Study Completion 2017-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: E. Wesley Ely, MD MPH, Principal Investigator — Tennessee Valley Healthcare System Nashville Campus, Nashville, TN
Locations (3):
- United States (3):
  - Tennessee Valley Healthcare System Nashville Campus, Nashville, TN, Nashville, Tennessee
  - VA Salt Lake City Health Care System, Salt Lake City, UT, Salt Lake City, Utah
  - VA Puget Sound Health Care System Seattle Division, Seattle, WA, Seattle, Washington

REFERENCES:
- [Background] Ely EW, Truman B, Shintani A, Thomason JW, Wheeler AP, Gordon S, Francis J, Speroff T, Gautam S, Margolin R, Sessler CN, Dittus RS, Bernard GR. Monitoring sedation status over time in ICU patients: reliability and validity of the Richmond Agitation-Sedation Scale (RASS). JAMA. 2003 Jun 11;289(22):2983-91. doi: 10.1001/jama.289.22.2983. PMID 12799407
- [Background] Ely EW, Inouye SK, Bernard GR, Gordon S, Francis J, May L, Truman B, Speroff T, Gautam S, Margolin R, Hart RP, Dittus R. Delirium in mechanically ventilated patients: validity and reliability of the confusion assessment method for the intensive care unit (CAM-ICU). JAMA. 2001 Dec 5;286(21):2703-10. doi: 10.1001/jama.286.21.2703. PMID 11730446
- [Background] Jackson JC, Gordon SM, Ely EW, Burger C, Hopkins RO. Research issues in the evaluation of cognitive impairment in intensive care unit survivors. Intensive Care Med. 2004 Nov;30(11):2009-16. doi: 10.1007/s00134-004-2422-2. Epub 2004 Sep 15. PMID 15372146
- [Background] Jackson JC, Gordon SM, Hart RP, Hopkins RO, Ely EW. The association between delirium and cognitive decline: a review of the empirical literature. Neuropsychol Rev. 2004 Jun;14(2):87-98. doi: 10.1023/b:nerv.0000028080.39602.17. PMID 15264710
- [Background] Ely EW, Wheeler AP, Thompson BT, Ancukiewicz M, Steinberg KP, Bernard GR. Recovery rate and prognosis in older persons who develop acute lung injury and the acute respiratory distress syndrome. Ann Intern Med. 2002 Jan 1;136(1):25-36. PMID 11777361
- [Background] Ely EW, Evans GW, Haponik EF. Mechanical ventilation in a cohort of elderly patients admitted to an intensive care unit. Ann Intern Med. 1999 Jul 20;131(2):96-104. doi: 10.7326/0003-4819-131-2-199907200-00004. PMID 10419447
- [Background] Hopkins RO, Weaver LK, Pope D, Orme JF, Bigler ED, Larson-LOHR V. Neuropsychological sequelae and impaired health status in survivors of severe acute respiratory distress syndrome. Am J Respir Crit Care Med. 1999 Jul;160(1):50-6. doi: 10.1164/ajrccm.160.1.9708059. PMID 10390379
- [Background] Ely EW, Margolin R, Francis J, May L, Truman B, Dittus R, Speroff T, Gautam S, Bernard GR, Inouye SK. Evaluation of delirium in critically ill patients: validation of the Confusion Assessment Method for the Intensive Care Unit (CAM-ICU). Crit Care Med. 2001 Jul;29(7):1370-9. doi: 10.1097/00003246-200107000-00012. PMID 11445689
- [Background] Ely EW, Gautam S, Margolin R, Francis J, May L, Speroff T, Truman B, Dittus R, Bernard R, Inouye SK. The impact of delirium in the intensive care unit on hospital length of stay. Intensive Care Med. 2001 Dec;27(12):1892-900. doi: 10.1007/s00134-001-1132-2. Epub 2001 Nov 8. PMID 11797025
- [Background] Ely EW, Shintani A, Truman B, Speroff T, Gordon SM, Harrell FE Jr, Inouye SK, Bernard GR, Dittus RS. Delirium as a predictor of mortality in mechanically ventilated patients in the intensive care unit. JAMA. 2004 Apr 14;291(14):1753-62. doi: 10.1001/jama.291.14.1753. PMID 15082703
- [Derived] Hughes CG, Hayhurst CJ, Pandharipande PP, Shotwell MS, Feng X, Wilson JE, Brummel NE, Girard TD, Jackson JC, Ely EW, Patel MB. Association of Delirium during Critical Illness With Mortality: Multicenter Prospective Cohort Study. Anesth Analg. 2021 Nov 1;133(5):1152-1161. doi: 10.1213/ANE.0000000000005544. PMID 33929361
- [Derived] Brummel NE, Bell SP, Girard TD, Pandharipande PP, Jackson JC, Morandi A, Thompson JL, Chandrasekhar R, Bernard GR, Dittus RS, Gill TM, Ely EW. Frailty and Subsequent Disability and Mortality among Patients with Critical Illness. Am J Respir Crit Care Med. 2017 Jul 1;196(1):64-72. doi: 10.1164/rccm.201605-0939OC. PMID 27922747
- See also: Click here for more information about this study: MIND-ICU Study: Delirium and Dementia in Veterans Surviving ICU Care — http://www.icudelirium.org